CLINICAL TRIAL: NCT02982369
Title: The Effects of Vertebral Manipulation and Pain Education in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Catarina Federal University (Other)
Responsible Party: Principal Investigator, Marcelo Anderson Bracht, Principal Investigator, Santa Catarina Federal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBracht; U1111-1190-4280 (Other: World Health Organization (WHO))
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Spinal Manipulation (Experimental): High-velocity and low-amplitude (HVLA) manipulation techniques to the cervical and thoracic region and pain education.
  The subjects will receive the treatment twice a week, for four weeks, totaling eight sessions, with an average duration of 30 minutes.
  Interventions: Other: Spinal Manipulation; Other: Pain Education
- Pain Education (Sham Comparator): Pain education and a simulation of spinal manipulation (sham), involving manual contact over the cervical and thoracic region totaling 10 minutes.
  The subjects will receive the treatment twice a week, for four weeks, totaling eight sessions, with an average duration of 30 minutes.
  Interventions: Other: Pain Education; Other: Sham

INTERVENTIONS:
Other: Spinal Manipulation — High-velocity and low-amplitude (HVLA) manipulation techniques to the cervical and thoracic region
  Other Names: Vertebral Manipulation
  Arms: Spinal Manipulation
Other: Pain Education — Subjects will receive pain education based in biopsychosocial approach
  Other Names: Pain Neuroscience Education
Other: Sham — A simulation of spinal manipulation (sham), involving manual contact over the cervical and thoracic region totaling 10 minutes.
  Arms: Pain Education

SUMMARY:
This study aims to investigate the effects of vertebral manipulation and pain education on subjects with neck pain. For this purpose, 90 subjects who present chronic neck pain will be selected and allocated randomly into 2 groups: vertebral manipulation group and pain education group.

ELIGIBILITY:
Inclusion Criteria:

* Main complaint of Neck Pain for at least six (6) months;
* Score of at least 10 points in NDI (Neck Disability Index);
* Pain and / or restriction of cervical movements;
* Pain reported at least 3 points on the NPRS (Numeric Pain Rating Scale);
* The definition of the term Neck Pain follows the classification of TFNP.

Exclusion Criteria:

* Previous history of rheumatic disease, cervical myelopathy, tumors, vertebrobasilar insufficiency, central or peripheral neurological disorders;
* History of major trauma, fracture or surgery in the neck, shoulder and/or upper limb;
* Signs of nerve root compression as important muscle weakness affecting the upper limbs, reduction, loss or increase of biceps and triceps reflexes, decreased sensation in the dermatomes of the upper limb;
* Red flags contraindicating spinal manipulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks after randomization
  Intensity of pain will be measured by the numeric pain rating scale (NPRS)

SECONDARY OUTCOMES:
Cytokines | 4 weeks after randomization
  Level of concentration of pro and anti-inflammatory cytokines
Pressure Pain Threshold | 4 weeks and 3 months after randomization
  Pressure pain Threshold will be measured with a digital algometer
Disability | 4 weeks and 3 months after randomization
  Disability will be measured by the Neck Disability Index (NDI)
Fear Avoidance Beliefs | 4 weeks and 3 months after randomization
  Fear Avoidance will be measured by the Fear Avoidance Beliefs Questionnaire (FABQ)
Health-related Quality of Life | 4 weeks and 3 months after randomization
  Quality of Life will be measured by the 12-Item Health Survey (SF-12)
Kinesiophobia | 4 weeks and 3 months after randomization
  Kinesiophobia will be measured byTampa Scale for Kinesiophobia
Pain Intensity | 3 months after randomization
  Intensity of pain will be measured by the numeric pain rating scale (NPRS)

CONTACTS AND LOCATIONS:
Overall Officials: Adair R Soares dos Santos, PhD, Study Director — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Florianópolis, Santa Catarina, Brazil